CLINICAL TRIAL: NCT02972489
Title: On-line 3-dimensional Optical Frequency Domain Imaging to Optimize Bifurcation Stenting Using UltiMaster Stent: OPTIMUM Study
Brief Title: Using 3D Imaging to Optimize Bifurcation Stenting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Increase Co., Ltd. (Industry)
Collaborators: Fujita Health University (Other); Erasmus Medical Center (Other); Terumo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTI001
Record Dates: First submitted 2016-11-14; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Artery Disease; Bifurcation Lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D OFDI guidance arm (Experimental): Bifurcation percutaneous coronary intervention (PCI) optimized by online-3D OFDI during and after procedure
  Interventions: Device: 3D OFDI guidance arm
- Angio guidance arm (Active Comparator): Bifurcation percutaneous coronary intervention (PCI) guided by angiography
  Interventions: Device: Angio guidance arm

INTERVENTIONS:
Device: 3D OFDI guidance arm — Subjects randomized to 3D-guidance arm will undergo optical frequency domain imaging (OFDI) assessment in the main vessel after re-wiring into the jailed side branch following stent implantation. If the position of the wire is not located in the optimal cell, further attempts to redirect the wire to the optimal cell will be performed, with subsequent OFDI acquisitions to confirm position in 2D and off-line 3D reconstruction. After procedure, OFDI is performed in the main branch.
  Arms: 3D OFDI guidance arm
Device: Angio guidance arm — In angiography-guidance group, wire recrossing into the side branch will be performed using conventional fluoroscopic/angiographic guidance. After finishing the procedure, OFDI is performed in the main branch but the results will be blinded to the operators.
  Arms: Angio guidance arm

SUMMARY:
The primary purpose of this study is to determine whether bifurcation stenting guided by on-line three-dimensional optical frequency domain imaging (3D-OFDI) is superior to that with angiographic guidance by measuring incomplete stent apposition (ISA) in the bifurcation segment.

DETAILED DESCRIPTION:
The recently developed optical frequency domain imaging (OFDI) can provide high quality resolution images of the coronary arteries. This new imaging system enhances the understanding of complex coronary lesions and the complex interaction between coronary devices and vessels by assembling/compiling 2-dimensional cross sections.

This 3-dimensional reconstruction with strut segmentation becomes possible on-line in the TERUMO OFDI console with 3-dimensional imaging software, which enables stent enhancement and 3D reconstruction within one minute. This "real time" 3D OFDI will promote the utilisation of 3-dimensional assessment in the treatment of bifurcation lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age and signed Informed Consent
2. Subject has coronary artery disease involving a bifurcation with objective evidence of ischemia including patients with chronic stable angina, silent ischemia and non-ST segment elevation acute coronary syndrome (NSTE-ACS)
3. Subject is appropriate to be treated by PCI according to the local practice (operator's judgment or heart team decision)
4. Patients' residence is in the area covered by the hospital
5. Patients with angiographically significant stenosis (>50 % by visual assessment) in de novo, native, previously unstented bifurcation lesion(s) including left main lesion, which is in operator's opinion appropriate to be treated by PCI with a single stent strategy
6. The size of main vessel matches available Ultimaster stent sizes (<4.0 mm, and 2.0 mm by visual assessment)
7. The size of side branch is >2.0mm in diameter by visual assessment
8. The sidebranch is treatable with a sidebranch fenestration and/or kissing balloon

Exclusion Criteria:

1. Pregnancy
2. Patients with ST elevation myocardial infarction
3. Known intolerance to aspirin, clopidogrel, heparin, cobalt chromium, sirolimus, contrast material
4. Known thrombocytopenia (platelet count< 100,000/mm3)
5. Cardiogenic Shock
6. Significant comorbidities precluding clinical follow-up (as judged by investigators)
7. Major planned surgery that requires discontinuation of dual antiplatelet therapy
8. History of stenting in the target bifurcation lesion
9. Renal insufficiency (GFR/MDRD <45 ml/min), which precludes in operator's opinion contrast injection during repeat OFDI pullback
10. Severely tortuous or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in sub-optimal optical frequency domain imaging (OFDI) or excessive risk of complication to place an OFDI catheter
11. Target lesion reference vessel diameter (RVD) < 2.25 and > 4 mm
12. Other: Patient is judged inappropriate by the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of malapposed struts | at time of bifurcation PCI surgery
  Percentage of malapposed struts assessed by OFDI in bifurcation segment of main vessel

SECONDARY OUTCOMES:
Incidence of fulfilling optimal recrossing criteria on 3D-OFDI | at time of bifurcation PCI surgery
  Measured as a percentage
Incomplete stent apposition (ISA) area (mm²) | at time of bifurcation PCI surgery
Minimum lumen area (mm²) | at time of bifurcation PCI surgery
Mean lumen area (mm²) | at time of bifurcation PCI surgery
Minimum stent area (mm²) | at time of bifurcation PCI surgery
Mean stent area (mm²) | at time of bifurcation PCI surgery
Mean protrusion area (mm²) | at time of bifurcation PCI surgery
Maximum protrusion area (mm²) | at time of bifurcation PCI surgery
Minimum flow area (mm²) | at time of bifurcation PCI surgery
Mean flow area (mm²) | at time of bifurcation PCI surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yoshinobu Onuma, Principal Investigator — Fujita Health University/Erasmus University Medical Center
Locations (2):
- Fujita Health University, Toyoake, Aichi-ken, Japan
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lassen JF, Holm NR, Stankovic G, Lefevre T, Chieffo A, Hildick-Smith D, Pan M, Darremont O, Albiero R, Ferenc M, Louvard Y. Percutaneous coronary intervention for coronary bifurcation disease: consensus from the first 10 years of the European Bifurcation Club meetings. EuroIntervention. 2014 Sep;10(5):545-60. doi: 10.4244/EIJV10I5A97. PMID 25256198
- [Background] Foin N, Torii R, Alegria E, Sen S, Petraco R, Nijjer S, Ghione M, Davies JE, Di Mario C. Location of side branch access critically affects results in bifurcation stenting: Insights from bench modeling and computational flow simulation. Int J Cardiol. 2013 Oct 9;168(4):3623-8. doi: 10.1016/j.ijcard.2013.05.036. Epub 2013 May 25. PMID 23714592
- [Background] Alegria-Barrero E, Foin N, Chan PH, Syrseloudis D, Lindsay AC, Dimopolous K, Alonso-Gonzalez R, Viceconte N, De Silva R, Di Mario C. Optical coherence tomography for guidance of distal cell recrossing in bifurcation stenting: choosing the right cell matters. EuroIntervention. 2012 Jun 20;8(2):205-13. doi: 10.4244/EIJV8I2A34. PMID 22581489
- [Background] Okamura T, Onuma Y, Garcia-Garcia HM, Bruining N, Serruys PW. High-speed intracoronary optical frequency domain imaging: implications for three-dimensional reconstruction and quantitative analysis. EuroIntervention. 2012 Feb;7(10):1216-26. doi: 10.4244/EIJV7I10A194. PMID 22334321
- [Background] Okamura T, Onuma Y, Yamada J, Iqbal J, Tateishi H, Nao T, Oda T, Maeda T, Nakamura T, Miura T, Yano M, Serruys PW. 3D optical coherence tomography: new insights into the process of optimal rewiring of side branches during bifurcational stenting. EuroIntervention. 2014 Dec;10(8):907-15. doi: 10.4244/EIJV10I8A157. PMID 24531393
- [Derived] Onuma Y, Kogame N, Sotomi Y, Miyazaki Y, Asano T, Takahashi K, Kawashima H, Ono M, Katagiri Y, Kyono H, Nakatani S, Muramatsu T, Sharif F, Ozaki Y, Serruys PW, Okamura T; OPTIMUM Investigators. A Randomized Trial Evaluating Online 3-Dimensional Optical Frequency Domain Imaging-Guided Percutaneous Coronary Intervention in Bifurcation Lesions. Circ Cardiovasc Interv. 2020 Dec;13(12):e009183. doi: 10.1161/CIRCINTERVENTIONS.120.009183. Epub 2020 Dec 4. PMID 33272034
- [Derived] Miyazaki Y, Muramatsu T, Asano T, Katagiri Y, Sotomi Y, Nakatani S, Takahashi K, Kogame N, Higuchi Y, Ishikawa M, Kyono H, Yano M, Ozaki Y, Serruys PW, Okamura T, Onuma Y. Online three-dimensional OFDI-guided versus angiography-guided PCI in bifurcation lesions: design and rationale of the randomised OPTIMUM trial. EuroIntervention. 2021 Mar 19;16(16):1333-1341. doi: 10.4244/EIJ-D-18-00902. PMID 31289018